CLINICAL TRIAL: NCT03100890
Title: In-home Versus Hospital Preoperative Training for Patients Undergoing Total Knee Replacement
Acronym: home_ATR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Politècnic i Universitari la Fe de València (Unknown)
Responsible Party: Principal Investigator, Jose María Blasco Igual, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRE_ATR_home
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hospitals; Home Care Services

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Non-active comparator
- Balance-Proprioception (Hospital) (Active Comparator): Preoperative training (hospital)
  Interventions: Other: Preoperative training (hospital)
- Balance-Proprioception (Home) (Experimental): Preoperative training (home)
  Interventions: Other: Preoperative training (home)

INTERVENTIONS:
Other: Preoperative training (hospital) — Preoperative hospital training
  Arms: Balance-Proprioception (Hospital)
Other: Preoperative training (home) — Preoperative in-home training
  Arms: Balance-Proprioception (Home)

SUMMARY:
In this work the importance of the potentiation and recovery of the balance with a physiotherapeutic intervention that begins in the early preoperative phase is compared with the conventional postoperative rehabilitation. The objective is to evaluate the influence of a muscle enhancement protocol in which a specific work of balance is included, with the physical benefits that this entails for the evolution of the patient. It also seeks to verify if the teaching and recommendation of exercises at home as preparation and conditioning for the intervention of ATR is effective, and to what extent, compared to a guided training in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe knee osteoarthritis that have not been operated before of total knee replacement.
* The score in Berg scale must be greater than 21.
* The score of the Mini-Mental State Examination must be equal or greater than 20.
* Once the informed consent is read and explained, patients must accept and agree to participate in the study.

Exclusion Criteria:

* Post-surgical infection of the operated knee.
* Pathology of central origin (i.e. cerebellar) that could interfere with balance or strength
* Vestibular pathology that could interfere with balance

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Self-reported functionality assessment
Berg Balance Scale (BBS) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Overall state of balance. Balance among older people with impairment in balance function by assessing the performance of functional tasks from the total score achieved in the 14 items test

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Dynamic balance assessment. Also points at the risk of falling. Time of getting up from a chair, walk three meters, come back and sit again, measured in seconds
Knee Range of Mobility (ROM) | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Knee Range of Mobility (Flexion, Extension) in degree
Quadriceps Strength | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Electronic dynamometer in Newton
Euro Quality of Life 5 Dimension | change from baseline to the week before surgery, 2 and 6 weeks after surgery
  Quality of Life assessment

CONTACTS AND LOCATIONS:
Overall Officials: José M Blasco, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blasco JM, Igual-Camacho C, Roig-Casasus S. In-home versus hospital preoperative balance and proprioceptive training in patients undergoing TKR; rationale, design, and method of a randomized controlled trial. BMC Musculoskelet Disord. 2017 Dec 8;18(1):518. doi: 10.1186/s12891-017-1887-4. PMID 29221471